CLINICAL TRIAL: NCT06627075
Title: Feasibility of Surface Optical Guidance to Replace the Restraint Mask for External Radiotherapy of Head and Neck Cancer
Brief Title: Optical Surface Guidance for External Radiotherapy of Head and Neck Cancer
Acronym: SUGAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-4-74-003; 2023-A02324-41 (Registry Identifier: ID RCB)
Record Dates: First submitted 2024-09-25; First posted 2024-10-04 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-09

CONDITIONS: Otorhinolaryngeal Cancer
Keywords: Radiotherapy; Optical surface guidance
MeSH Terms: conditions — Otorhinolaryngologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surface Guided RadioTherapy without face mask (Experimental): Radiotherapy sessions will be carried out using the surface camera system, replacing the restraint mask.
  Self-assessment questionnaires will also be completed by healthcare professionals concerning the level of difficulty encountered during each SGRT session without mask.
  Skin side effects are recorded by the radiotherapist during weekly follow-up consultations.
  At the end of treatment, patients complete a patient experience questionnaire.
  Interventions: Procedure: Surface Guided RadioTherapy (SGRT) without mask

INTERVENTIONS:
Procedure: Surface Guided RadioTherapy (SGRT) without mask — Firstly, patients are positioned in a vacuum mattress that moulds their head, neck and shoulders for a reference scan.
  During the treatment sessions, patients are positioned according to the reference scan, using the surface camera system.
  Once the observed offsets have been applied, the patient's surface is captured. Treatment can then begin, with continuous monitoring of displacements by the surface camera system. Automatic beam interruption is provided during treatment in the event of motion detection exceeding the standard tolerance threshold (>3 mm).
  If the use of a thermoformed mask during your treatment prove necessary, for whatever reason, will not result in a halt to the research.
  Patients receive between 10 and a max of 35 radiotherapy sessions. The follow-up period begins after the last radiotherapy session, and patients are assessed at 4 or 6 weeks and at 3 months by a radiotherapist.

SUMMARY:
The goal of this clinical trial is to test the use of surface repositioning alone, without a restraint mask, during radiotherapy sessions for patients with head and neck cancer.

DETAILED DESCRIPTION:
In radiotherapy treatments for head and neck cancer, the use of a mask is recommended for patient immobilization. The mask completely covers the head and shoulders, ensuring reproducible positioning at every session. However, using a mask can be oppressive and anxiety-provoking for patients.

At the same time, technological developments have led us to use optical surface camera systems to position and monitor patients in the treatment room. In this way, if a movement exceeding the threshold is detected during a session, the treatment is automatically interrupted.

However, despite the use of the mask, movements are still possible underneath, and are not detected by the surface cameras.

The study's hypothesis is that the use of surface repositioning alone could guarantee reproducible treatment, as in combination with a thermoformed mask. In addition, eliminating the mask would mean greater comfort and improved quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients undergoing palliative or curative treatment for oro-rhino-laryngeal cancer
* Patients with an indication for radiotherapy treatment, with or without complementary treatment (chemotherapy, immunotherapy), with a number of sessions between 10 and 35
* Patients who have dated and signed an informed consent form

Exclusion Criteria:

* Patients with uncontrollable movements
* Patients under psychiatric care
* Patients who do not understand or read French
* Patients participating in an interventional study testing another medical intervention
* Patients under guardianship, curatorship, safeguard of justice or deprived of liberty
* Pregnant or breast-feeding women
* Patients without social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
Measurement patient displacement during surface-guided radiotherapy sessions | Through study completion, an average of 1 year
  Average length of linear translation vector during session (measured by surface cameras) over all sessions performed

CONTACTS AND LOCATIONS:
Overall Officials: Coralie Geffroy, Principal Investigator — Centre de Lutte contre le Cancer Eugène Marquis
Locations (1):
- Centre de Lutte contre le Cancer Eugène Marquis, Rennes, Brittany Region, France